CLINICAL TRIAL: NCT04633304
Title: A Single Arm sTudy to Evaluate the Effectiveness of EndoAVF in a Pre-dialysis Population
Brief Title: A Single Arm sTudy to Evaluate the Effectiveness of EndoAVF in a Pre-dialysis Population (STEP Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: California Institute of Renal Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STP-001
Record Dates: First submitted 2020-10-09; First posted 2020-11-18 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: CKD Stage 3; CKD Stage 4; CKD Stage 5
Keywords: CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: primary end point
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- AVF (Other): Single arm study using primary and secondary end points as comperators between subjects.
  Interventions: Device: EndoAVF System for endovascular AV fistula creation

INTERVENTIONS:
Device: EndoAVF System for endovascular AV fistula creation — AV fistula creation
  Other Names: WavelinQ™

SUMMARY:
This is an investigator-initiated post-marketing study that will evaluate use of the WaveLinQ system, a new and novel method of fistula creation using a percutaneous method in patients who require the creation of an arteriovenous fistula (AVF).

DETAILED DESCRIPTION:
This investigator-initiated post-marketing study will evaluate use of the WaveLinQ system, a new and novel method of fistula creation, which uses a percutaneous method to create an AVF. Thirty male and female subjects with CKD 3-5 and who are clinical indicated for arteriovenous fistula (AVF) creation will be enrolled using the WaveLinQ device. Eligibility confirmation will be confirmed during screening up to 28 days from the index procedure. Subjects who are eligible will undergo fistula creation per standard institutional technique (index/baseline) and be followed at least monthly for 6 months per their standard of care plan. Primary, clinical and functional patency will be observed throughout the trial in addition to other data collection points per protocol. The expected total duration of subject participation from screening until the end of study is up to 7 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female Age of at least 18 years
2. CKD 3 through 5 as measured by GFR 45 and under by MDRD equation on two separate occasions at least 3 months apart.
3. Provide written informed consent using a form that is approved by the Institutional Review Board (IRB) prior to collection of study data or performance of study procedures.
4. Currently not on hemodialysis.
5. Life expectancy of at least one year
6. Meets Anatomical Criteria for EndoAVF creation via pre-procedure Duplex or Venography Vascular anatomy suitable for creation of the AV fistula
7. Willing to comply with the specified follow-up evaluations

Exclusion Criteria:

1. Anatomical exclusion criteria met
2. Thought to need dialysis within 30 days.
3. The subject is in a hypercoagulable state.
4. The subject has known bleeding diathesis.
5. The subject has insufficient cardiac output to support a native fistula in the opinion of the investigator.
6. Known history of active intravenous drug abuse.
7. The subject has a known allergy or hypersensitivity to contrast media which cannot be adequately pre-medicated.
8. The subject has known adverse effects to sedation and/or anesthesia which cannot be adequately pre-medicated.
9. Evidence of active infection on the day of the index procedure (temperature of ≥ 38.0° Celsius and/ or WBC of ≥ 12,000 cells/ μL, if collected).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedure Success | Interval of time from access placement until any intervention is undertaken to maintain or re-establish patency - 6 weeks
  Successful endoAVF creation confirmed by intraprocedural angiography or duplex Ultrasound post procedure

SECONDARY OUTCOMES:
Physiologically mature endoAVF at 6 months | 6 months
  Percent of patients who did not require any intervention to be undertaken to maintain or re-establish patency

CONTACTS AND LOCATIONS:
Overall Officials: Osman Khawar, MD, Principal Investigator — California Institute of Renal Research
Locations (1):
- California Institute of Renal Research, Escondido, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones RG, Khawaja A, Tullett K, Inston NG. Early experience and observations in endovascular dialysis fistula re-intervention. J Vasc Access. 2020 Nov;21(6):818-825. doi: 10.1177/1129729819888374. Epub 2019 Dec 9. PMID 31814515
- [Background] Inston N, Khawaja A, Tullett K, Jones R. WavelinQ created arteriovenous fistulas versus surgical radiocephalic arteriovenous fistulas? A single-centre observational study. J Vasc Access. 2020 Sep;21(5):646-651. doi: 10.1177/1129729819897168. Epub 2020 Jan 2. PMID 31894716
- [Result] Lok CE, Rajan DK, Clement J, Kiaii M, Sidhu R, Thomson K, Buldo G, Dipchand C, Moist L, Sasal J; NEAT Investigators. Endovascular Proximal Forearm Arteriovenous Fistula for Hemodialysis Access: Results of the Prospective, Multicenter Novel Endovascular Access Trial (NEAT). Am J Kidney Dis. 2017 Oct;70(4):486-497. doi: 10.1053/j.ajkd.2017.03.026. Epub 2017 Jun 14. PMID 28624422
- [Result] Radosa CG, Radosa JC, Weiss N, Schmidt C, Werth S, Hofmockel T, Plodeck V, Gatzweiler C, Laniado M, Hoffmann RT. Endovascular Creation of an Arteriovenous Fistula (endoAVF) for Hemodialysis Access: First Results. Cardiovasc Intervent Radiol. 2017 Oct;40(10):1545-1551. doi: 10.1007/s00270-017-1750-x. Epub 2017 Aug 7. PMID 28785804
- [Result] Berland TL, Clement J, Griffin J, Westin GG, Ebner A. Endovascular Creation of Arteriovenous Fistulae for Hemodialysis Access with a 4 Fr Device: Clinical Experience from the EASE Study. Ann Vasc Surg. 2019 Oct;60:182-192. doi: 10.1016/j.avsg.2019.02.023. Epub 2019 May 8. PMID 31075457
- [Result] Zemela MS, Minami HR, Alvarez AC, Smeds MR. Real-World Usage of the WavelinQ EndoAVF System. Ann Vasc Surg. 2021 Jan;70:116-122. doi: 10.1016/j.avsg.2020.05.006. Epub 2020 May 15. PMID 32417285